CLINICAL TRIAL: NCT05769855
Title: A Phase 3, Multicenter, Randomized, Double-Blind, Parallel-Group, Active and Placebo Controlled Study to Evaluate the Efficacy and Safety of Local Administration of HR18034 for Postoperative Analgesia in Subjects Undergoing Hemorrhoidectomy
Brief Title: A Study of HR18034 for Postoperative Analgesia in Subjects Undergoing Hemorrhoidectomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Shanghai Hengrui Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HR18034-301
Record Dates: First submitted 2023-03-03; First posted 2023-03-15 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2023-02

CONDITIONS: Postsurgical Pain Management
MeSH Terms: interventions — Ropivacaine

STUDY DESIGN:
Intervention Model Description: HR18034 compared with active comparator and placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- HR18034 (Experimental)
  Interventions: Drug: HR18034
- ropivacaine HCl (Active Comparator)
  Interventions: Drug: ropivacaine HCl
- Sodium Chloride Physiological Solution (Placebo Comparator)
  Interventions: Drug: Sodium Chloride Physiological Solution

INTERVENTIONS:
Drug: HR18034 — HR18034 380mg
  Arms: HR18034
Drug: ropivacaine HCl — ropivacaine HCl 75mg.
  Arms: ropivacaine HCl
Drug: Sodium Chloride Physiological Solution — Sodium Chloride Physiological Solution 20ml
  Arms: Sodium Chloride Physiological Solution

SUMMARY:
The study is being conducted to evaluate the efficacy, and safety of HR18034 for postoperative analgesia in subjects undergoing hemorrhoidectomy.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide a written informed consent
2. Subjects requiring hemorrhoidectomy under subarachnoid anesthesia
3. 18 kg/m2 ≤ BMI ≤ 30 kg/m2
4. Conform to the ASA Physical Status Classification
5. Women of childbearing age have a negative pregnancy test and are not nursing

Exclusion Criteria:

1. Subjects with a history of myocardial infarction or unstable angina pectoris
2. Subjects with atrioventricular block or cardiac insufficiency
3. Subjects with a history of ischemic stroke or transient ischemic attack
4. Subjects with a history of mental illness and a history of cognitive impairment epilepsy
5. Subjects with concurrent painful physical condition that may affect postoperative pain assessment
6. Spinal or spinal lesions that were determined by the investigator to be unable to tolerate subarachnoid anesthesia
7. Subjects with a history of hemorrhoidectomy
8. Subjects with a history of constipation
9. Subjects with a history of perianal disease
10. Abnormal values in the laboratory
11. Subject with heart rate <50 or >100 beats per minute.
12. Subject with refractory hypertension
13. History of hypersensitivity or idiosyncratic reactions to amide-type local anesthetics, opioids, or other drugs that may used in study
14. History of prohibited drug use
15. Participants who may be affected by alcohol, or drug abstinence during the study period;
16. Participated in clinical trials of other drugs (received experimental drugs)
17. The inestigators determined that other conditions were inappropriate for participation in this clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 294 (Actual)
Dates: Start 2023-03-21 (Actual); Primary Completion 2023-10-30 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
AUC of Pain Intensity in rest state | 0~72 hours after administration
  Pain intensity will be evaluated using an 11-point (0-10) Numeric Pain Rating Scale (NPRS), with higher numbers indicating a higher pain intensity, administered over 72 hours.

SECONDARY OUTCOMES:
Proportion of subjects with Pain Rating Scale (NPRS)≥4 during dressing change | 0~72 hours after administration
Proportion of subjects with Pain Rating Scale (NPRS)≥4 during defecation | 0~72 hours after administration
AUC of Pain Intensity in rest state | 0~24 hours after administration
AUC of Pain Intensity in move state | 0~24 hours，0~72 hours after administration
Proportion of subjects who doesn't recive rescue analgesic | 0~72 hours after administration
Participant's satisfaction score for analgesia treatment | 72-hours
Investigator's satisfaction score for analgesia treatment | 72-hours

CONTACTS AND LOCATIONS:
Locations (1):
- The Third Xiangya Hospital of Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Undecided